CLINICAL TRIAL: NCT03499678
Title: Clinical Trials on Detection of Lung Cancer With Non-invasive Method Based on DNA Methylation of Circulated Tumor DNA, PBMC and T Cells
Brief Title: Lung Cancer Screening Using DNA Methylation Changes in Circulated Tumor and PBMC DNA
Status: Terminated | Type: Observational
Why Stopped: Encountered technical issues with blood plasma samples received from the hospital.
Sponsor: HKGepitherapeutics (Industry)
Collaborators: Kazakh Research Institute of Oncology & Radiology (Other)
Responsible Party: Sponsor
Other Study IDs: HKG-KZ-LNG-102
Record Dates: First submitted 2018-03-28; First posted 2018-04-17 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Lung Cancer; Lung Cancer, Nonsmall Cell; Lung Cancer, Small Cell
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA extracted from PBMC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung Cancer: Small cell lung cancers (SCLC) and non-small cell lung cancers (NSCLC)
- Control: Age and sex matched control individuals

SUMMARY:
A central challenge in the fight against lung cancers is how to detect disease in a noninvasive manner before it is detectable by imaging methods. Although inroads have been made with more sensitive imaging techniques for earlier detection of breast and lung cancers, these techniques are limited by the size of lesion that could be detected. Alternatively, several blood proteomic biomarkers have been proposed but none offer as of yet sufficient predictive power. Consequently, effective non-invasive tools as prognostic indicators and biomarkers of lung cancer is urgently needed.

The purpose of this study is to develop and test non-invasive biomarkers based on methylation changes in PBMC and circulated tumor DNA in lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed lung cancer

Exclusion Criteria:

* Pregnant women
* Minors (subjects less than 18 years of age)
* Prisoners
* Patients with known infectious disease, such as human immunodeficiency virus (HIV), tuberculosis (TB), or hepatitis B, C
* Patients having other than one cancer
* Subjects unable to consent for themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be assigned an ID that will be kept confidential according to hospital regulations. IDs will be randomized so that identity will not be revealed except to the approved hospital personnel. Methylation data will be returned to the hospital for follow up of progression of disease and for assessing early prediction of progression of lung cancer and will be entered into the data base. Other clinical follow up data will be entered into the electronic data base. All data will be captured in case report form.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
DNA methylation of circulated tumor and PBMC DNA and its Correlation to Development and prediction of lung cancer | 6 months to 1 year
  The outcome is the methylation score, which combines the weighted methylation values of four CpGs. A threshold methylation score that differentiates between control and cancer individuals will be calculated from the training set of 100 patients.
  The model will be provided to the researchers:
  Methylation score=CG1*b1+CG2*b2+ CG3*b3+ CG4*b4 + e
  CG1 is the methylation value of the first CG b1 is the regression coefficient for the first CG and "e" equals the intercept. Investigators will develop the regression coefficient and intercept as well as the DNA methylation values for each patient for each CG. Investigators will first compute the polygenic methylation score for each patient. Then based on the computer threshold based on the training cohort will call the samples as lung cancer or not.

CONTACTS AND LOCATIONS:
Locations (1):
- Kazakh Institute of Oncology and Radiology, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided